CLINICAL TRIAL: NCT01185158
Title: A Phase II Study of 250-mg ZD1839 Monotherapy in Recurrent or Metastatic or Both Recurrent and Metastatic Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11588A
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer
Keywords: Larynx; Lip; Oral Cavity and Pharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases; Lymphoid Interstitial Pneumonia | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZD1839 (IRESSA) 250mg (Experimental): ZD1839(IRESSA) 250mg orally (po) daily
  Interventions: Drug: ZD1839 (IRESSA)

INTERVENTIONS:
Drug: ZD1839 (IRESSA) — ZD1839: 250mg/day po or via g-tube Q 24 hours

SUMMARY:
The purpose of this study is to find out what effects (good and bad) ZD1839 has on one's squamous cell head and neck cancer. The research is being done because currently no effective treatment exists for metastatic (spread of cancer cells from one area of the body to another) or recurrent squamous cell cancer of the head and neck. The purpose of this study is to find out if ZD1839 can shrink tumors or cause tumors to stop growing for a period of time.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck incurable by surgery or radiation
* Patients must have measurable disease, defined as at least on e lesion that can be accurately measured in the one dimension (longer diameter to be recorded) as greater then or equal to 20mm with conventional techniques or as greater than or equal to 10mm with computed tomograpy (CT) scan.

Therapeutic history that includes the Following:

* No prior EGFR-based therapy for recurrent disease
* No chemotherapy or irradiation with the 28-day period preceding entry to the study
* Eastern Cooperative Oncology Group (ECOG)performance Status 0-2 (kamofsky >59%)

Patients must have normal organ and marrow function as defined below:

* leukocytes >3,000ml
* absolute neutrophil count 1,500/ml
* platelets 100,000/ml
* total bilirubin within normal institutional limits
* AST(SGOT)ALT(SGPT) <2.5 X institutional upper limits of normal
* Creatinine <1.5

Exclusion Criteria:

* Other coexisting malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical in situ.
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, ketoconazole, erythromycin, clarithromycin, atorvastatin, cimetidine, ametidine, amitriptyline, imipramine, verpamil, tamoxifen, chlorpromazine, amiodorone, chloroquine, St. John's Wort
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy
* Incomplete healing from previous oncologic or other major surgery Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compound of similar chemical or biologic composition to ZD 1839
* Uncontrolled intercurrent illness
* Pregnancy or breast feeding (women of child -bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2002-05; Primary Completion 2004-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To assess the activity of 250mg of ZD1839 administered as a single agent to patients with recurrent or metastatic or both recurrent and metastatic head and neck cancer. | 2 -5 years

SECONDARY OUTCOMES:
To demonstrate the effectiveness of ZD 1839 as an inhibitor of epithelial growth factor (EGFR) phosphorylation, MAP kinase activation, and vascular endothelial growth (VEGF) secretion in metastatic head and neck cancer. | 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, M.D., Principal Investigator — The Univesity of Chicago Medical Center
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- See also: The University of Chicago Comprehensive Cancer Center Web page — http://uccrc.uchicago.edu